CLINICAL TRIAL: NCT04440293
Title: Effects of Basic Body Awareness Therapy on Pain, Balance and Proprioceptive Sense in Patients With Chronic Neck Pain
Brief Title: Effects of Basic Body Awareness Therapy on Patients With Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: KaratayUKY
Record Dates: First submitted 2020-06-16; First posted 2020-06-19 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Neck Pain; Proprioceptive Disorders; Balance; Distorted
Keywords: neck pain; proprioception; balance; body awareness; exercise
MeSH Terms: conditions — Neck Pain; Somatosensory Disorders; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group BBAT / CT (Experimental): Group BBAT / CT started treatment with BBAT and received 2 days a week for 6 weeks. After the interval of 5-week, group BBAT / CT was treated with CT twice a week for 6 weeks.
  Interventions: Other: BBAT; Other: CT
- Group CT / BBAT (Experimental): Group CT / BBAT started treatment with CT and received 2 days a week for 6 weeks. After the interval of 5-week, group CT / BBAT was treated with BBAT twice a week for 6 weeks.
  Interventions: Other: BBAT; Other: CT

INTERVENTIONS:
Other: BBAT — The BBAT was applied by a trained and certified physiotherapist in this area for about an hour, two days a week, as a group therapy. The BBAT program includes movements related to daily activities such as lying, sitting, standing and walking. BBAT focuses on basic movement principles such as postural stability, energy adjustment in movements, comfortable breathing and coordination.
Other: CT — The CT program was applied two days a week for about an hour. The CT program includes active range of motion (ROM) exercises, stretching, isometric and resistant strengthening, posture exercises and relaxation training.

SUMMARY:
The aim of this study was to compare the effects of Basic Body Awareness Therapy (BBAT) and conventional therapies (CT) on pain, balance and proprioceptive sensation of cervical region in patients with chronic neck pain. As a cross-over study, patients were divided into BBAT / CT (n=17) and CT / BBAT (n=18) groups. BBAT program has been implemented to patients within group BBAT / CT two days a week for 6 weeks while group CT / BBAT received the CT program during the same period. After the interval of 5-week, group BBAT / CT was treated with CT and group CT / BBAT was treated with BBAT. Pain severity with; Visual Analogue Scale (VAS), disability level with; Neck Disability Index (NDI), cervical proprioception with; Cervical Range of Motion Deluxe (CROM) device, balance with; Computerized Dynamic Posturography were evaluated. The evaluations were conducted before and after the first and second treatment.

DETAILED DESCRIPTION:
Chronic neck pain is a common musculoskeletal disease that affects many people at some point in life.Its prevalence in the general population varies between 30-50% and is more common in women over 50 years old.The cervical area is an important body part due to the sensorial receptors of the muscles and joints as well as central and reflexes connections with visual, vestibular, and postural control systems.Numerous sensorimotor disorders have been detected in patients with chronic neck pain.Some patients with neck pain have impaired proprioceptive sensation and postural control.Pain can affect presynaptic inhibition of muscle afferents and modulation of proprioceptive muscle spindles, causing prolonged delays.These changes may result in decreased muscle control and increased postural release.Different updated and conventional therapy (CT) methods are used for the treatment of neck pain. Mobilization of soft tissue and joint, stabilization techniques, cervical collars, relaxation training, strengthening exercises, and posture arrangement by body awareness are common therapeutic modalities. Basic Body Awareness Therapy (BBAT) is a method used by physiotherapists to increase patient awareness and control posture.The method is increasingly used in the treatment of painful conditions related to the chronic musculoskeletal system.However, there are not enough studies in the literature examining the effects of proprioceptive senses and postural control in patients with chronic neck pain. The aim of this study is to compare the effects of BBAT and conventional treatments (CT) on pain, balance and proprioceptive sensation of the cervical region in patients with chronic neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 or over,
* Having neck pain for more than 3 months,
* Having neck problems that do not cause neurological deficits

Exclusion Criteria:

* History of cervical vertebra fracture or spinal tumor,
* Those diagnosed with cervical dystonia,
* Whiplash-related disorders,
* Those diagnosed with vertigo, fibromyalgia, or rheumatoid arthritis,
* The presence of inflammatory disease or infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-04-02 (Actual); Study Completion 2018-05-16 (Actual)

PRIMARY OUTCOMES:
Balance | at the beginning of treatments
  The balance assessed by the Sensorial Organization Test (SOT) in the Computerized Dynamic Posturography device.The results of the SOT are calculated according to anterior-posterior sways. A balance score ranging from 0 to 100 is achieved, where 0 indicates loss of balance and 100 indicates excellent stability.
Balance | 6 weeks later
  The balance assessed by the Sensorial Organization Test (SOT) in the Computerized Dynamic Posturography device.The results of the SOT are calculated according to anterior-posterior sways. A balance score ranging from 0 to 100 is achieved, where 0 indicates loss of balance and 100 indicates excellent stability.
Balance | 11 weeks later
  The balance assessed by the Sensorial Organization Test (SOT) in the Computerized Dynamic Posturography device.The results of the SOT are calculated according to anterior-posterior sways. A balance score ranging from 0 to 100 is achieved, where 0 indicates loss of balance and 100 indicates excellent stability.
Balance | 17 weeks later
  The balance assessed by the Sensorial Organization Test (SOT) in the Computerized Dynamic Posturography device.The results of the SOT are calculated according to anterior-posterior sways. A balance score ranging from 0 to 100 is achieved, where 0 indicates loss of balance and 100 indicates excellent stability.
Neck proprioception | at the beginning of treatments
  Proprioceptive sensation was evaluated using the Cervical Range of Motion Deluxe (CROM, Deluxe Performance Attainment Associates, Lindstrom, Minnesota, USA) device.Joint position error and deflection angles of the head in all 3 planes were measured with CROM device.
Neck proprioception | 6 weeks later
  Proprioceptive sensation was evaluated using the Cervical Range of Motion Deluxe (CROM, Deluxe Performance Attainment Associates, Lindstrom, Minnesota, USA) device.Joint position error and deflection angles of the head in all 3 planes were measured with CROM device.
Neck proprioception | 11 weeks later
  Proprioceptive sensation was evaluated using the Cervical Range of Motion Deluxe (CROM, Deluxe Performance Attainment Associates, Lindstrom, Minnesota, USA) device.Joint position error and deflection angles of the head in all 3 planes were measured with CROM device.
Neck proprioception | 17 weeks later
  Proprioceptive sensation was evaluated using the Cervical Range of Motion Deluxe (CROM, Deluxe Performance Attainment Associates, Lindstrom, Minnesota, USA) device.Joint position error and deflection angles of the head in all 3 planes were measured with CROM device.

SECONDARY OUTCOMES:
Pain severity | at the beginning of treatments
  Visual Analogue Scale (VAS) was used to determine the severity of pain in the patients with neck pain. Patients were asked to indicate their pain levels on a scale of 0-10 cm. The value "0" indicates no pain while the value "10" indicates unbearable pain.
Pain severity | 6 weeks later
  Visual Analogue Scale (VAS) was used to determine the severity of pain in the patients with neck pain. Patients were asked to indicate their pain levels on a scale of 0-10 cm. The value "0" indicates no pain while the value "10" indicates unbearable pain.
Pain severity | 11 weeks later
  Visual Analogue Scale (VAS) was used to determine the severity of pain in the patients with neck pain. Patients were asked to indicate their pain levels on a scale of 0-10 cm. The value "0" indicates no pain while the value "10" indicates unbearable pain.
Pain severity | 17 weeks later
  Visual Analogue Scale (VAS) was used to determine the severity of pain in the patients with neck pain. Patients were asked to indicate their pain levels on a scale of 0-10 cm. The value "0" indicates no pain while the value "10" indicates unbearable pain.
Neck disability level | at the beginning of treatments
  The Neck Disability Index was used to determine the patients' neck disability levels. There are ten sections of the scale that question the severity of pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation, consisting of 6 questions. Item scores range from 0 (no disability) to 5 (total disability).
Neck disability level | 6 weeks later
  The Neck Disability Index was used to determine the patients' neck disability levels. There are ten sections of the scale that question the severity of pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation, consisting of 6 questions. Item scores range from 0 (no disability) to 5 (total disability).
Neck disability level | 11 weeks later
  The Neck Disability Index was used to determine the patients' neck disability levels. There are ten sections of the scale that question the severity of pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation, consisting of 6 questions. Item scores range from 0 (no disability) to 5 (total disability).
Neck disability level | 17 weeks later
  The Neck Disability Index was used to determine the patients' neck disability levels. There are ten sections of the scale that question the severity of pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation, consisting of 6 questions. Item scores range from 0 (no disability) to 5 (total disability).

CONTACTS AND LOCATIONS:
Overall Officials: Kamil Yılmaz, 1, Principal Investigator — KTO Karatay University
Locations (1):
- KTO Karatay University, Konya, Turkey (Türkiye)